CLINICAL TRIAL: NCT01249703
Title: The Early Diagnosis and Warning Role of Erectile Dysfunction:a Multi-institutional Clinical Study.
Brief Title: The Early Diagnosis and Warning Role of Erectile Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Chunhua Deng, Department of Urology
Other Study IDs: Chunhua Deng
Record Dates: First submitted 2010-11-29; First posted 2010-11-30 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2008-01

CONDITIONS: Erectile Dysfunction; Endothelial Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: Yes

SUMMARY:
1. Find the early diagnostic markers of erectile dysfunction;
2. Study the warning role of ED in some diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Male and at least 18 years of age.
2. Provide signed informed consent.
3. Have a history of erectile dysfunction (ED: defined as a consistent change in the quality of erection that adversely affects the subject's satisfaction with sexual intercourse) .
4. Have a stable monogamous relationship with a female partner. To some subjects with poor sexual experience, re-evaluation would be conducted after a 4-weeks sex education.
5. Make at least four sexual intercourse attempts with the female sexual study partner during the 4-week therapeutic period without medication.
6. Agree not to use any other ED treatment for at least 4 weeks.

Exclusion Criteria:

1. severe diseases (such as congestive heart failure, arrhythmia, significant renal or hepatic dysfunction and anemia);
2. Had clinically noteworthy penile deformities, pelvic surgery or trauma of perineal region;
3. Had received long-term pharmacotherapy (including antioxidant agents, vitamins and traditional Chinese drugs).
4. An addiction problem (with a history of injection or administration of opium, poppy, heroin, hemp, morphine, cocaine, caffeine, ketamine and meperidine etc.)

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: men with erectile dysfunction healthy men general male population
Sampling Method: Probability Sample
Enrollment: 150000 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-10 (Actual); Study Completion 2020-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Chunhua Deng, MD, PhD, Principal Investigator — Department of Urology
Locations (1):
- The First Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China